CLINICAL TRIAL: NCT05065476
Title: Assessing the Impact of Isha Kriya Meditation on Anxiety and Depression - a Pilot Study
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Balachundhar Subramaniam, Professor of Anesthesia, Beth Israel Deaconess Medical Center
Other Study IDs: 2021P000359
Record Dates: First submitted 2021-09-23; First posted 2021-10-04 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Anxiety; Depression
Keywords: meditation; anxiety; depression; Isha Kriya
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: Participants signed up for the webinar will be learning and practicing the "Isha Kriya" practice (meditation for beginners) taught by the Isha Foundation.

SUMMARY:
This study aims to assess the impact of Isha Kriya, a freely available guided meditation, on mental health - specifically anxiety and depression.

DETAILED DESCRIPTION:
In 2019, over 15% of the population experienced symptoms of anxiety. This was highest amongst 18-29-year-olds. Amongst these adults, 9.5% experienced mild, 3.4% experienced moderate, and 2.7% experienced severe symptoms of anxiety. About 1 in 6 adults is expected to suffer from depression at some point in their lives. Due to the pandemic, rates of anxiety and depression increased significantly. In December 2020, 42% of people surveyed by the US Census Bureau had symptoms associated with anxiety or depression. This is compared to 11% of adults having similar symptoms from Jan-June 2019. The rapidly diminishing mental health in the general population, especially since the COVID-19 pandemic, has raised the concern for an emerging new pandemic: the mental health pandemic. Mental health leaders and organizations are urging the federal and state authorities to make mental health a top priority and allocate resources to areas including early identification and prevention, establishing integrated health and mental health care to ensure "whole-person" well-being, assuring evidence-based standards of prevention, treatment and care.

Meditation has been shown to be effective in reducing symptoms associated with anxiety and depression. A recent study using a meditation called Isha Kriya showed improved perceived stress amongst operating room professionals in one sitting. Isha Kriya is a simple meditation practice (15minutes) that can be done by anyone over 12 years of age. It is offered free globally via in-person sessions, online webinars, and online videos. A meditation which is available electronically and freely could be an attractive option to include in prevention and treatment strategies for anxiety and depression. Furthermore, such intervention is easily scalable and accessible to everyone with access to the internet and if found effective, can be a valuable resource for addressing disparities in access to mental health resources in minority and underserved populations. This study aims to assess the effectiveness of this meditation on reducing symptoms associated with anxiety and depression over 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* Interest in Isha Kriya

Exclusion Criteria:

* Low English proficiency
* Not currently residing in United States

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from a pool of healthy volunteers who sign up for a webinar where they learn the "Isha Kriya" practice. Isha Foundation has developed the Isha Kriya practice and conducts online Isha Kriya webinars (Meditation for Beginners). This webinar is routinely conducted by Isha Foundation.
Sampling Method: Non-Probability Sample
Enrollment: 267 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Compliance | Changes from baseline to 6 weeks
  The weekly compliance questionnaire is a tool which helps the participants to keep a track of their activities each week. This enables the study team to measure compliance and protocol adherence by the participants by collecting information on their routine activity practiced and its frequency.

SECONDARY OUTCOMES:
PROMIS - Anxiety Short Form | Changes from baseline to 6 weeks
  PROMIS - Anxiety Short Form1 is an 8 item validated instrument that assesses severity of anxiety. Participants are asked on a scale of 1 (Never) to 5 (Always) on the frequency of occurrence of each negative experience. Overall score is computed based on sum from individual responses.
Center for Epidemiological Studies Depression Scale (CES-D-10) | Changes from baseline to 6 weeks
  PROMIS - Anxiety Short Form is an 8 item validated instrument that assesses severity of anxiety.
  Participants are asked on a scale of 1 (Never) to 5 (Always) on the frequency of occurrence of each negative experience. Overall score is computed based on sum from individual responses.

CONTACTS AND LOCATIONS:
Overall Officials: Sepideh Hariri, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Terlizzi EP, Villarroel MA. Symptoms of Generalized Anxiety Disorder Among Adults: United States, 2019. NCHS Data Brief. 2020 Sep;(378):1-8. PMID 33054928
- [Background] Kessler RC, Berglund P, Demler O, Jin R, Merikangas KR, Walters EE. Lifetime prevalence and age-of-onset distributions of DSM-IV disorders in the National Comorbidity Survey Replication. Arch Gen Psychiatry. 2005 Jun;62(6):593-602. doi: 10.1001/archpsyc.62.6.593. PMID 15939837
- [Background] Abbott A. COVID's mental-health toll: how scientists are tracking a surge in depression. Nature. 2021 Feb;590(7845):194-195. doi: 10.1038/d41586-021-00175-z. No abstract available. PMID 33536600
- [Background] Saeed SA, Cunningham K, Bloch RM. Depression and Anxiety Disorders: Benefits of Exercise, Yoga, and Meditation. Am Fam Physician. 2019 May 15;99(10):620-627. PMID 31083878
- [Background] Saeed SA, Antonacci DJ, Bloch RM. Exercise, yoga, and meditation for depressive and anxiety disorders. Am Fam Physician. 2010 Apr 15;81(8):981-6. PMID 20387774
- [Background] Gonzalez-Valero G, Zurita-Ortega F, Ubago-Jimenez JL, Puertas-Molero P. Use of Meditation and Cognitive Behavioral Therapies for the Treatment of Stress, Depression and Anxiety in Students. A Systematic Review and Meta-Analysis. Int J Environ Res Public Health. 2019 Nov 10;16(22):4394. doi: 10.3390/ijerph16224394. PMID 31717682
- [Background] Rangasamy V, Thampi Susheela A, Mueller A, F H Chang T, Sadhasivam S, Subramaniam B. The effect of a one-time 15-minute guided meditation (Isha Kriya) on stress and mood disturbances among operating room professionals: a prospective interventional pilot study. F1000Res. 2019 Mar 26;8:335. doi: 10.12688/f1000research.18446.1. eCollection 2019. PMID 32665843
- [Derived] Hariri S, Vishnubhotla RV, Reed PU, Rayapuraju A, Orui H, Balachundhar P, Sadhasivam S, Subramaniam B. Online guided meditation training (Isha Kriya) improves self-reported symptoms of anxiety and depression within 2 weeks of practice-An observational study. Front Psychiatry. 2022 Sep 23;13:944973. doi: 10.3389/fpsyt.2022.944973. eCollection 2022. PMID 36213913
- See also: Related Info — http://www.apa.org/news/press/releases/2020/12/mental-health-organizations